CLINICAL TRIAL: NCT07117058
Title: Validation of a Rapid Screening Tool for Anxiety-depressive Disorders in Children, Adolescents and Young Adults Treated in Oncology. Multicenter Study. Short Title: HARMONY-Tool
Brief Title: Validation of a Rapid Screening Tool for Anxiety-depressive Disorders in Children, Adolescents and Young Adults Treated in Oncology. Multicenter Study.
Acronym: HARMONY-Tool
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 23CH131; 2024-A02404-43 (Other: ANSM)
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Generalized Anxiety; Introspective & Anxiety-Prone Patient; Depression, Anxiety; Survivors of Childhood Cancer
Keywords: anxiety symptoms; childhood cancer; screening; psychological complication
MeSH Terms: conditions — Generalized Anxiety Disorder; Depression; Anxiety Disorders; Neoplasms | interventions — Early Detection of Cancer

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- 7-10 years old group: Develop and validate, using a psychometric method, a rapid screening tool for anxiety-depressive disorders in children cured of childhood cancer.
  Interventions: Diagnostic Test: New rapid screening tool for anxiety and depressive disorders; Diagnostic Test: SCARED-R-51 (Screen for Child Anxiety Related Emotional Disorders-Revised)
- 11-14 years old group: Develop and validate, using a psychometric method, a rapid screening tool for anxiety-depressive disorders in adolescents cured of childhood cancer.
  Interventions: Diagnostic Test: New rapid screening tool for anxiety and depressive disorders; Diagnostic Test: SCARED-R-51 (Screen for Child Anxiety Related Emotional Disorders-Revised)
- 15-25 years old group: Develop and validate, using a psychometric method, a rapid screening tool for anxiety-depressive disorders in young adults cured of childhood cancer.
  Interventions: Diagnostic Test: New rapid screening tool for anxiety and depressive disorders; Diagnostic Test: HADS (Hospital Anxiety and Depression Scale)

INTERVENTIONS:
Diagnostic Test: New rapid screening tool for anxiety and depressive disorders — New rapid screening tool for anxiety and depressive disorders completed by patient during a regular follow-up consultation
Diagnostic Test: SCARED-R-51 (Screen for Child Anxiety Related Emotional Disorders-Revised) — Questionnaire completed by patient during a regular follow-up consultation : ONLY for patients 7-14 years old.
  Groups: 11-14 years old group; 7-10 years old group
Diagnostic Test: HADS (Hospital Anxiety and Depression Scale) — Questionnaire completed by patient during a regular follow-up consultation : ONLY for patients 15-25 years old.
  Groups: 15-25 years old group

SUMMARY:
In France today, it is estimated that one in every 850 people aged between 20 and 45 is a childhood cancer survivor (CCS), equivalent to around 40,000 to 50,000 people. Some descriptive studies have established that the diagnosis and treatment of cancer can affect psychological health. A French study published by our team in 2015 and 2020 showed that in adulthood, 40% of CCS had anxiety symptoms, a rate significantly higher than that of the general French population (25%). However, although there are validated scales for screening children for psychological disorders (anxiety, depression, etc.), there is no rapid screening tool that can be used routinely by an oncologist during consultations. So, the study aims to develop and validate a short test, which could easily be carried out systematically during follow-up consultations after childhood cancer. It would make it possible to identify people with no psychological complications and, conversely, those in whom further investigation, based on the classic reference scales for assessing psychological disorders, would be relevant.

DETAILED DESCRIPTION:
The aim of the HARMONY-Tool study is to develop and validate, using a psychometric method, a rapid screening tool for anxiety-depressive disorders in children, adolescents and young adults cured of childhood cancer.

ELIGIBILITY:
Inclusion Criteria

* Patients diagnosed with pediatric cancer before the age of 18,
* Patient whose intensive treatment had ended at least 3 months prior to inclusion,
* Patients considered to be in complete remission by the doctor responsible for their treatment,
* Patient affiliated to or entitled under a social security scheme,
* Patient having received informed information about the study OR the holder(s) of parental authority having received informed information about the study in the case of minors.

Exclusion Criteria

* Refusal to participate expressed by the patient or minor,
* Patients whose cancer has relapsed or progressed,
* Pregnant women, women in labor, breast-feeding mothers,
* Persons deprived of their liberty, hospitalized without consent, hospitalized for purposes other than those of the research,
* Adults under legal protection (guardianship) or unable to express their consent.

Ages: 7 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients diagnosed with pediatric cancer before the age of 18, whose intensive treatment had ended at least 3 months prior to inclusion and considered to be in complete remission by the doctor responsible for their treatment,
Sampling Method: Non-Probability Sample
Enrollment: 545 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
New rapid screening tool for anxiety-depressive disorders | At inclusion
  This tools is under construction.
  Items development of this tool is following 3 steps :
  1. Identification of dimensions and generation of items : a combination of a deductive method (literature review) and an inductive method (questioning individuals) are used to identify the various dimensions relevant to the early assessment of anxiety and depressive disorders and generate the corresponding items.
  2. Content validity : the expert judges method to confirm, supplement, or reduce the initial selection of items are used
  3. Response options for content validity : binary response options for questions that are unambiguous are used.
  This tool will contain a maximum of 7 questions for children aged 6 to 10, 8 questions for adolescents aged 11 to 14 (in particular because of an additional question on the use of addictive substances) and 10 questions for the 15-25 age group (with the possibility of finer dimensions)
SCARED-R-51 (Screen for Child Anxiety Related Emotional Disorders-Revised) | At inclusion
  Only for 7-14 years old
HADS (Hospital Anxiety and Depression Scale) | At inclusion
  Only 15-25 years old

CONTACTS AND LOCATIONS:
Overall Officials: CLAIRE BERGER, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (5):
- France (5):
  - Centre Hospitalier Universitaire, Grenoble
  - IHOP, Lyon
  - Centre Hospitalier Universitaire, Rouen
  - CHU de Saint-Etienne, Saint-Etienne
  - Centre Hospitalier Universitaire, Tours

IPD SHARING:
Plan to Share IPD: Undecided